CLINICAL TRIAL: NCT04726007
Title: Management of Therapeutic Antithrombotic in Patients With VTE After Stroke and Hemorrhagic Tendency
Brief Title: Management of TA in VaS-Patients and HT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Wang JingWen-1
Record Dates: First submitted 2021-01-20; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2020-12

CONDITIONS: VTE After Stroke
MeSH Terms: interventions — Fibrinolytic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antithrombotic Agents — Antithrombotic agents include anticoagulants, antiplatelet drugs, thrombolytic drugs.

SUMMARY:
Stroke is an independent risk factor for venous thrombosis (VTE), which leads to a significant increase in the mortality and disability rate after stroke. For patients with high risk factors for VTE such as advanced age, paralysis, infection, dehydration, etc., the incidence of death and disability is higher. Studies have shown that the incidence of deep vein thrombosis in bedridden ischemic stroke patients is about 20%, and the incidence of pulmonary embolism is about 2%, and causes 10% of post-stroke deaths. In order to prevent the occurrence of VTE, the American Heart Association, the American Stroke Association, the Cerebrovascular Disease Group of the Neurology Branch of the Chinese Medical Association, etc. pointed out in the guidelines that heparin or low molecular weight heparin should be used for stroke patients with "restricted mobility" or "incapable mobility" to prevent VTE. For patients with evidence of thrombosis or symptoms of DVT, antithrombotic therapy should be initiated immediately. Paradoxically, ischemic stroke significantly increases the risk of cerebral hemorrhage. Besides There is an increased risk of primary intracerebral hemorrhage (ICH) associated with aspirin or antiplatelet agent monotherapy and it is difficult to achieve a balance between preventing blood clots and reducing the risk of bleeding complications. In addition, stroke patients are elderly and have speech and intellectual impairment, and the non-specific symptoms and signs of intracranial hemorrhage caused by improper antithrombotic therapy make the rate of misdiagnosis and missed diagnosis extremely high. Therefore, clarifying the clinical characteristics of stroke patients with VTE and launching targeted interventions to effectively balance the risk of anti-thrombosis and bleeding have become the key to improving the prognosis of patients.

This study is based on real-world data to study the bleeding risk and antithrombotic treatment options in VaS (1) the risk factors associated with hemorrhage in patients with VTE after stroke; and (2) the characteristics and pharmacotherapeutics regimen of high-risk populations with VTE after stroke; and(3) the Optimal antithrombotic treatment regimen for patients with VTE after stroke, including the timing of starting and stopping the antithrombotic treatment, selection of varieties, dosage, and course of treatment, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with VTE after stroke
* Use at least one antithrombotic drug

Exclusion Criteria:

* Case information is incomplete
* Non-spontaneous cerebral hemorrhage
* Suffer from serious blood system disease
* Do not accept follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We integrated pooled individual patient data of consecutive VaS patients treated at a single center (Departments of Neurology) in China from 1 January 2008 until 31 December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Complications during hospital stay in patients with VTE after stroke | Through study completion, an average of 2 weeks.
  Bleeding is defined as intracranial hemorrhage and non-intracranial hemorrhage, and thrombosis is defined as aggravated or new thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jingwen Wang, Study Director — The First Affiliated Hospital of the Air Force Medical University
Locations (1):
- The First Affiliated Hospital of the Air Force Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes